CLINICAL TRIAL: NCT02717299
Title: Making Sense Out of Total Knee Sensor Assisted Technology: A Randomized Control Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: TriHealth Inc. (Other)
Collaborators: Orthosensor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-053
Record Dates: First submitted 2016-03-15; First posted 2016-03-23 (Estimated); Last update posted 2020-05-04 (Actual); Status verified 2019-04

CONDITIONS: Arthroplasty, Replacement, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sensor Guided Tissue Balancing (Experimental): Patients in this group will have the Verasense trial sensor device inserted, and the data collected electronically. The surgeon will use this data to intraoperatively align the knee according to the indications of the data.
  Interventions: Device: Verasense
- Surgeon Guided Tissue Balancing (Placebo Comparator): Patients in this group will have the Verasense trial sensor device inserted, and the data collected electronically. The computer displaying the data will be turned away from the surgeon, so that he is not able to use the sensor data, and must balance the knee with feel and visual estimation of balance.
  Interventions: Device: Verasense

INTERVENTIONS:
Device: Verasense — Verasense will collect balancing data on all patients in this trial.

SUMMARY:
The purpose of this study is to compare the patient reported outcome measures of total knee replacement patients who received intra operative sensor guided technique for soft tissue balancing to a group of patients who receive surgeon guided soft tissue balancing.

DETAILED DESCRIPTION:
This study will compare a group of total knee arthroplasty patients who receive sensor guidance technology for soft tissue balancing intra operatively to a group of patients who receive surgeon guided soft tissue balancing. Patients will be randomized to either the experimental group with the sensor guided technology or the control group which is the surgeon guided technique and current standard of care. All patients will have the sensor placed intra operatively so that measurements can be captured and recorded however, the measurements for the patients who are not in the sensor guided group will not be revealed to the surgeon. The information will be gathered for post enrollment data analysis only. The patients measurements in the sensor guided group will be revealed to the surgeon and the surgeon will use this information in order to help guide soft tissue balancing for optimal alignment intra operatively. Patients will be followed for 1 year post operatively. Patient reported outcomes measures such as KSS, KOOS, PROMIS PF CAT, EQ-5D and UCLA activity will be collected preoperatively and at 3 months, 6 months, and 12 months. Post-operative Likert scale patient satisfaction scores will also be collected. All outcomes will be scored and compared to determine significance.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing primary unilateral total knee arthroplasty for osteoarthritis, avascular necrosis, inflammatory arthropathy, or post traumatic arthritis.
* Patients able to understand study intent, and agree to study participation.
* Patients receiving Smith and Nephew Journey II total knee implant system.

Exclusion Criteria:

* Patients with previous ipsilateral knee ligament surgery.
* Patients with orthopaedic and medical co-morbidities that would thwart postoperative recovery such as extra-articular pathology with referred pain to the knee (spinal stenosis, neuropathy, ipsilateral hip disease), severe knee deformity.
* Untreated Osteoarthritis
* BMI > 40
* ASA class > III
* History of drug or alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2015-11 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2021-04-08 (Estimated)

PRIMARY OUTCOMES:
Patient Satisfaction | Surgery to 12 months post-operative
  Overall Patient Satisfaction will be reported through various surveys.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Snyder, MD, Principal Investigator — TriHealth Inc.
Locations (1):
- Good Samarian Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Yes, Orthosensor receives the data collected.